CLINICAL TRIAL: NCT06521671
Title: Evaluation of Femoral Neck Fracture Migration After Internal Fixation With an Angle Stable Implant Compared With Gold Standard Cannulated Cancellous Screws in Young Adults: Study Protocol for a Clinical RCT Using Radiostereometric Analysis
Brief Title: Evaluation of Fracture Migration After Internal Fixation of Femoral Neck Fractures in Younger Adults: A Clinical RCT Using RSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Region of Southern Denmark (Other); Swemac Innovation AB (Unknown); Gødstrup Hospital (Other)
Responsible Party: Principal Investigator, Michaela Manalili Hansen, Medical Doctor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2401073
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Femoral Neck Fractures; Internal Fixation; Complications; Hip Fractures
Keywords: femoral neck fracture; radiostereometric analysis; hip fracture; internal fixation
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Randomisation groups will be kept blinded during statical analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynaloc (Experimental): Randomisation
  Interventions: Device: Dynaloc implant
- Cannulated cancellous screws (Active Comparator): Randomisation
  Interventions: Device: Cannulated cancellous screws
- Sliding hip screw (Active Comparator): Prospective cohort
  Interventions: Device: Sliding hip screw

INTERVENTIONS:
Device: Dynaloc implant — Internal fixation with Dynaloc implant
  Arms: Dynaloc
Device: Cannulated cancellous screws — Internal fixation with two or three cannulated cancellous screws
  Arms: Cannulated cancellous screws
Device: Sliding hip screw — Internal fixation with a sliding hip screw
  Arms: Sliding hip screw

SUMMARY:
The goal of the clinical trial is to compare different surgical methods for internal fixation of femoral neck fractures in younger adults.

The main question it aims to answer is:

Is internal fixation with the novel implant consisting of three angle stable screws locked together by a plate equal to internal fixation with cancellous screws or a sliding hip screw in younger adults under 65 years of age in terms of fracture migration?

The study will examine how stable the fracture remains during healing. This will be measured by assessing how much the fracture moves after surgery using a highly precise imaging method called radiostereometric analysis (RSA). The study will also record complications and evaluate pain, health related quality of life, and hip function over time.

The participants will be treated with either a novel angle stable implant (Dynaloc), cannulated cancellous screws or sliding hip screw and followed up at 6 weeks, 12 weeks, 6 months and 12 months. Recruitment will continue until 75 participants, 25 in each group, have completed the 12-week follow-up for the primary outcome.

DETAILED DESCRIPTION:
Objective The overall purpose of the study is to assess internal fixation methods for femoral neck fractures in adults under 65 years of age. The primary objective is to compare fracture migration following internal fixation with a novel angle-stable implant (Dynaloc, Swemac) and cannulated cancellous screws (CCS), using fracture migration as the primary outcome.

In addition, a cohort of patients treated with a sliding hip screw (SHS) as part of standard care will be included to provide an additional basis for comparison.

Dynaloc, CCS, and SHS are all CE-marked medical devices used in accordance with the manufacturers' intended use.

Trial design The study is designed as a multicentre, single-blinded randomised controlled trial with radiostereometric analysis (RSA), including an additional prospective cohort.

Patients undergoing internal fixation with Dynaloc or CCS will be randomised, while patients treated with a sliding hip screw will be followed as a separate cohort using the same imaging and follow-up protocol.

Interventions Eligible patients will be randomised to internal fixation with either three CCS or the Dynaloc implant.

Patients who do not undergo randomisation and are treated with SHS as standard care may be included in a prospective cohort and followed according to the study protocol.

All surgical procedures will be performed according to the manufacturers' surgical techniques and instructions for use.

Sample size calculation The primary outcome is shortening of the femoral neck at 12 weeks. A clinically relevant difference is defined as femoral neck shortening greater than 5 mm. Femoral neck shortening in patients treated with CCS is expected to be 5.3 mm (SD 4.5 mm) at 6 weeks, and no further clinically relevant shortening is expected between 6 and 12 weeks.

Using a power of 0.9, a significance level of 0.05, and assuming a maximum femoral neck shortening of 1 mm in the Dynaloc group compared with 5.3 mm (SD 4.5 mm) in the CCS group, a total sample size of 50 randomised patients (25 per group) is required.

In addition, a cohort of 25 patients treated with a sliding hip screw will be included for comparative purposes.

Inclusion will continue until all 50 randomised patients and all 25 cohort patients have completed the 12-week follow-up for the primary outcome. Due to the rarity of femoral neck fractures in this age group, up to approximately 20% additional patients may be included to ensure complete 12-week follow-up.

Randomization/allocation After informed consent is obtained, eligible patients will be enrolled and entered into an electronic database. Patients will be randomised to either CCS or Dynaloc using block randomisation with block sizes of 4 and 6. Randomisation will be stratified by Garden classification (Garden 1-2 vs. 3-4) to account for fracture displacement and by hospital of admission.

The operating surgeon will contact a central coordinator to perform the randomisation prior to surgery and will therefore know the allocated implant before entering the operating theatre.

Blinding Participants and care providers will be blinded to the allocated implant. A standardised description of the surgical procedure will be used. Treatment allocation will remain blinded during statistical analyses.

Data Collection Project staff will collect clinical data, CT scans, and radiostereometric X-rays and perform image analyses using AutoRSA. Screening will be conducted by the admitting physician. Baseline data will be collected during admission and entered directly into REDCap by project personnel.

Patient-reported outcome questionnaires will be distributed electronically via REDCap, with responses automatically uploaded to the database. Follow-up visits will take place in the outpatient clinic, where project personnel will complete and verify data entry.

Statistical methods Treatment groups will remain blinded during statistical analyses. Data distribution will be assessed and results presented accordingly. Continuous outcomes will be analysed using linear mixed-effects models, and categorical variables will be compared using χ² or Fisher's exact tests, as appropriate.

A p-value of <0.05 will be considered statistically significant. Postoperative complication rates will be defined as the combined incidence of complications and reoperations. Mortality will be analysed using Cox regression. Statistical analyses and graphical presentation will be performed using STATA 18 (StataCorp).

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck fracture (DS720)
* Age 18-64 years
* Ability to speak and read Danish
* Willingness to participate

Exclusion Criteria:

* Pathological, basicervical or transcervical fracture
* Clinical Frailty Scale ≥5, indicating mild to severe frailty prior to the fracture
* Cognitive impairment that hinders informed consent
* Previous fracture in the ipsilateral femur
* Patients who are unwilling or incapable of following post-operative care instructions.
* Comorbidities making the participant ineligible for internal fixation such as:

  * Material sensitivity, documented or suspected
  * Active or suspected latent infection, sepsis or marked local inflammation in or around the surgical area
  * Compromised vascularity, inadequate skin or neurovascular status
  * Compromised bone stock that cannot provide adequate support and/or fixation of the device due to disease, infection or prior implantation
  * Other physical, mental, medical or surgical conditions that would preclude the potential benefit of surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Static fracture migration | 12 weeks
  Static non-weight bearing fracture migration in a supine set-up

SECONDARY OUTCOMES:
Static fracture migration | 6 weeks
  Static non-weight bearing fracture migration in a supine set-up
New mobility score | Baseline, 6 weeks, 12 weeks
  Assessment of gait. 0-9 points
Modified Harris Hip Score | Baseline, 6 weeks, 12 weeks
  Measure of hip dysfunction. <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
EQ-5D-5L | Baseline, 6 weeks, 12 weeks
  Health related Quality of Life
Pain VRS | Baseline, 6 weeks, 12 weeks
  Pain verbal rating scale 0-10
Reoperation | 0-12 weeks
  Any secondary operation
Complication | 0-12 weeks
  Any complication (non-union, avascular necrosis of the femoral head, fixation failure)
Mortality | 0-12 weeks
  Death

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Regional Hospital Gødstrup, Gødstrup
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen MM, Petersen ET, Gundtoft PH, Jensen J, Stilling M, Ding M, Viberg B. Evaluation of femoral neck fracture migration after internal fixation with an angle stable implant compared with gold standard cannulated cancellous screws in young adults: study protocol for a clinical RCT using radiostereometric analysis. Trials. 2026 Feb 7. doi: 10.1186/s13063-026-09497-7. Online ahead of print. PMID 41652608